CLINICAL TRIAL: NCT03900975
Title: Analyses of the Outcome of a Treatment of Vulvar Paget Disease
Brief Title: Vulvar Paget Disease
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2018/1164
Record Dates: First submitted 2018-12-14; First posted 2019-04-03 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Vulvar Paget's Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vulvar Paget Disease: Women with vulvar paget disease

SUMMARY:
In this study only women with vulvar paget disease will be included and will be analysed retrospectively. Vulvar paget disease patients are frequently treated with surgical resection of the affected tissue. During a surgical treatment surgical margins are frequently positive. Recidives are seen frequently after surgical treatment or the development of other pathologies such as vulvar carcinoma. In this study the outcome of the vulvar paget disease will be analysed and compared between the participants. It's primary goal is to create a better view on the outcome and the prognosis to prevent e.g. complications in the future.

DETAILED DESCRIPTION:
In this study only women with vulvar paget disease will be included and will be analysed retrospectively. Vulvar paget disease patients are frequently treated with surgical resection of the affected tissue. During a surgical treatment surgical margins are frequently positive. Recidives are seen frequently after surgical treatment or the development of other pathologies such as vulvar carcinoma. In this study the outcome of the vulvar paget disease will be analysed and compared between the participants. It's primary goal is to create a better view on the outcome and the prognosis to prevent e.g. complications in the future.

All the information of the patients will be gathered retrospectively from their medical file , after they gave their consent.

ELIGIBILITY:
Inclusion Criteria:

* Vulvar Paget disease

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women will be included
Study Population: Women with vulvar paget disease
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of complications after the treatment of vulvar Paget disease | Max. 10 years after treatment
  Number of complications after treatment
Type of complications after the treatment of vulvar Paget disease | Max. 10 years after treatment
  Type of complications after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium